CLINICAL TRIAL: NCT01462435
Title: A Phase 3, Randomized, Double-Blind, Multiple-Dose, Parallel-Group, Active- and Placebo-Controlled Study of Diclofenac [Test] Capsules for the Treatment of Acute Postoperative Pain After Bunionectomy
Brief Title: Study of Diclofenac Capsules to Treat Pain Following Bunionectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Iroko Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DIC3-08-04
Record Dates: First submitted 2011-10-26; First posted 2011-10-31 (Estimated); Results first posted 2013-12-19 (Estimated); Last update posted 2014-02-04 (Estimated); Status verified 2014-01

CONDITIONS: Other Acute Postoperative Pain
MeSH Terms: interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Diclofenac Test (lower dose) (Experimental)
  Interventions: Drug: Diclofenac Test (lower dose)
- Diclofenac Test (upper dose) (Experimental)
  Interventions: Drug: Diclofenac Test (upper dose)
- Celecoxib (Active Comparator)
  Interventions: Drug: Celecoxib
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diclofenac Test (lower dose) — Capsules
  Arms: Diclofenac Test (lower dose)
Drug: Diclofenac Test (upper dose) — Capsules
  Arms: Diclofenac Test (upper dose)
Drug: Celecoxib — 200 mg Capsules
  Arms: Celecoxib
Drug: Placebo — Capsules
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether Diclofenac [Test] Capsules are safe and effective for the treatment of bunionectomy pain.

ELIGIBILITY:
Inclusion Criteria:

* Patient is male or female between 18 and 65 years of age
* For women of child-bearing potential: a woman who is not pregnant and not nursing, and who is practicing an acceptable method of birth control
* Has undergone primary, unilateral, first metatarsal bunionectomy with no additional collateral procedures
* Patient must be willing to stay at the study site ≥ 72 hours

Exclusion Criteria:

* Patient has hypersensitivity, allergy, or clinically significant intolerance to any medications to be used in the study, or related drugs
* Patient has a current disease or history of a disease that will impact the study or the patient's well-being
* Patient has used or intends to use any of the medications that are prohibited by the protocol
* Patient has a history of drug or alcohol abuse or dependence, or patient has a positive urine drug screen or alcohol breathalyzer test
* Patient has taken another investigational drug within 30 days prior to screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2011-10; Primary Completion 2012-02 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Golf, DPM, Principal Investigator — Premier Research Group Limited; Ira Gottlieb, DPM, Principal Investigator — Chesapeake Research Group, LLC; Kyle Patrick, DO, Principal Investigator — Premier Research Group Limited; S. Thomas Schiffgen, DPM, Principal Investigator — Premier Research Group Limited
Locations (4):
- United States (4):
  - Premier Research Group Limited, Phoenix, Arizona
  - Chesapeake Research Group, LLC, Pasadena, Maryland
  - Premier Research Group Limited, Austin, Texas
  - Premier Research Group Limited, Salt Lake City, Utah

REFERENCES:
- [Derived] Argoff C, McCarberg B, Gudin J, Nalamachu S, Young C. SoluMatrix(R) Diclofenac: Sustained Opioid-Sparing Effects in a Phase 3 Study in Patients with Postoperative Pain. Pain Med. 2016 Oct;17(10):1933-1941. doi: 10.1093/pm/pnw012. Epub 2016 Mar 19. PMID 26995799

RESULTS

PARTICIPANT FLOW:
Groups:
- Celecoxib: Celecoxib : 200 mg Capsules
- Diclofenac Test (Lower Dose): Diclofenac Test (lower dose) : Capsules
- Diclofenac Test (Upper Dose): Diclofenac Test (upper dose) : Capsules
- Placebo: Placebo : Capsules
Period: Overall Study
Arm/Group | Celecoxib | Diclofenac Test (Lower Dose) | Diclofenac Test (Upper Dose) | Placebo
Started | 106 | 109 | 107 | 106
Completed | 105 | 109 | 106 | 101
Not Completed | 1 | 0 | 1 | 5
Not completed — Lack of Efficacy | 1 | 0 | 0 | 3
Not completed — Physician Decision | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Celecoxib | Diclofenac Test (Lower Dose) | Diclofenac Test (Upper Dose) | Placebo | Total
Number analyzed (Participants) | 106 | 109 | 107 | 106 | 428
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (11.9) | 39.4 (11.7) | 39.3 (11.8) | 39.9 (12.6) | 39.7 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 94 | 89 | 92 | 371
  Male | 10 | 15 | 18 | 14 | 57
Region of Enrollment [Number; unit: participants]
  United States | 106 | 109 | 107 | 106 | 428

OUTCOME MEASURES:

1. Primary Outcome: The Time-Weighted Summed Pain Intensity Difference Measured Using the 100-mm Visual Analogue Scale From 0 to 48 Hours After Trial Entry (VASSPID-48), ANCOVA Model.
Description: The pain intensity is assessed using a visual analogue scale (VAS), which is a horizontal line 100 mm in length. Subjects mark the VAS with a single vertical line to indicate their current pain level, with 0 mm representing "No Pain" and 100 mm representing "Worst Possible Pain".
  The VAS summed pain intensity difference (VASSPID) is calculated as the sum of the pain intensity difference values at each follow-up time point (difference between the starting pain intensity and the pain intensity at the given assessment time) multiplied by the amount of time (in hours) since the prior assessment.
Time Frame: 0 - 48 hours
Population: Intent-to-Treat Population
Measure: Mean (Standard Deviation); unit: mm*hour
Arm/Group | Celecoxib | Diclofenac Test (Lower Dose) | Diclofenac Test (Upper Dose) | Placebo
Number analyzed (Participants) | 106 | 109 | 107 | 106
mm*hour | 390.468 (925.1) | 392.954 (937.0) | 524.315 (1146.1) | 76.887 (340.6)
Statistical Analysis 1: Comparison: Diclofenac Test (Upper Dose) vs Placebo; Test type: Superiority or Other; p < 0.001, ANCOVA; Difference in Least Squares Mean = 446.946, 95% CI 2-sided [206.567 to 687.324], Standard Error of Mean 122.2935
Statistical Analysis 2: Comparison: Diclofenac Test (Lower Dose) vs Placebo; Test type: Superiority or Other; p = 0.010, ANCOVA; Difference in Least Squares Mean = 316.145, 95% CI 2-sided [77.136 to 555.155], Standard Error of Mean 121.5971
Statistical Analysis 3: Comparison: Celecoxib vs Placebo; Test type: Superiority or Other; p = 0.011, ANCOVA; Difference in Least Squares Mean = 313.119, 95% CI 2-sided [72.202 to 554.037], Standard Error of Mean 122.5676

2. Secondary Outcome: VASSPID-4. The Time-Weighted Summed Pain Intensity Difference Measured Using the 100-mm Visual Analogue Scale (VASSPID) From 0 to 4 Hours After Trial Entry.
Description: as for outcome 1
Time Frame: 0 - 4 hours
Measure: Mean (Standard Deviation); unit: mm*hour
Arm/Group | Celecoxib | Diclofenac Test (Lower Dose) | Diclofenac Test (Upper Dose) | Placebo
Number analyzed (Participants) | 106 | 109 | 107 | 106
mm*hour | 25.109 (62.9) | 27.450 (64.9) | 31.568 (68.6) | 14.406 (53.5)
Statistical Analysis 1: Comparison: Diclofenac Test (Upper Dose) vs Placebo; Test type: Superiority or Other; p = 0.043, t-test, 2 sided
Statistical Analysis 2: Comparison: Diclofenac Test (Lower Dose) vs Placebo; Test type: Superiority or Other; p = 0.109, t-test, 2 sided
Statistical Analysis 3: Comparison: Celecoxib vs Placebo; Test type: Superiority or Other; p = 0.183, t-test, 2 sided

3. Secondary Outcome: VASSPID-8. The Time-Weighted Summed Pain Intensity Difference Measured Using the 100-mm Visual Analogue Scale (VASSPID) From 0 to 8 Hours After Trial Entry.
Description: as for outcome 1
Time Frame: 0 - 8 hours
Measure: Mean (Standard Deviation); unit: mm*hour
Arm/Group | Celecoxib | Diclofenac Test (Lower Dose) | Diclofenac Test (Upper Dose) | Placebo
Number analyzed (Participants) | 106 | 109 | 107 | 106
mm*hour | 51.675 (122.4) | 56.404 (132.6) | 64.689 (138.5) | 23.151 (84.9)
Statistical Analysis 1: Comparison: Diclofenac Test (Upper Dose) vs Placebo; Test type: Superiority or Other; p = 0.009, t-test, 2 sided
Statistical Analysis 2: Comparison: Diclofenac Test (Lower Dose) vs Placebo; Test type: Superiority or Other; p = 0.029, t-test, 2 sided
Statistical Analysis 3: Comparison: Celecoxib vs Placebo; Test type: Superiority or Other; p = 0.050, t-test, 2 sided

4. Secondary Outcome: VASSPID-24. The Time-Weighted Summed Pain Intensity Difference Measured Using the 100-mm Visual Analogue Scale (VASSPID) From 0 to 24 Hours After Trial Entry.
Description: as for outcome 1
Time Frame: 0 - 24 hours
Measure: Mean (Standard Deviation); unit: mm*hour
Arm/Group | Celecoxib | Diclofenac Test (Lower Dose) | Diclofenac Test (Upper Dose) | Placebo
Number analyzed (Participants) | 106 | 109 | 107 | 106
mm*hour | 170.845 (393.0) | 177.101 (418.3) | 230.708 (499.9) | 48.811 (186.5)
Statistical Analysis 1: Comparison: Diclofenac Test (Upper Dose) vs Placebo; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Diclofenac Test (Lower Dose) vs Placebo; Test type: Superiority or Other; p = 0.004, t-test, 2 sided
Statistical Analysis 3: Comparison: Celecoxib vs Placebo; Test type: Superiority or Other; p = 0.004, t-test, 2 sided

5. Secondary Outcome: Total Pain Relief (TOTPAR) Over 0 to 4 Hours. TOTPAR-4.
Description: Pain relief was assessed using a 5-point categorical scale at all assessment time points after time 0. Subjects were asked "How much relief have you had since your starting pain?" with response choices of none = 0, a little = 1, some = 2, a lot = 3, and complete = 4.
  The Total Pain Relief (TOTPAR) score for a given time interval is calculated as the sum of the pain relief scores at each follow-up time point (as recorded on the categorical pain relief scale) over that interval multiplied by the amount of time (in hours) since the prior assessment. In this way individual scores covering a longer time period were given more weight.The minimum theoretical score is 0 units, which represent no relief from pain (score of 0 on categorical scale) at all time points after time 0. The maximum theoretical score is 16 units, which represents complete relief from pain (score of 4 on a categorical scale) at all time points after time 0.
Time Frame: 0 - 4 hours
Measure: Mean (Standard Deviation); unit: units on a scale*hour
Arm/Group | Celecoxib | Diclofenac Test (Lower Dose) | Diclofenac Test (Upper Dose) | Placebo
Number analyzed (Participants) | 106 | 109 | 107 | 106
units on a scale*hour | 2.226 (3.5) | 2.112 (3.5) | 2.530 (3.6) | 1.387 (2.7)
Statistical Analysis 1: Comparison: Diclofenac Test (Upper Dose) vs Placebo; Test type: Superiority or Other; p = 0.009, t-test, 2 sided
Statistical Analysis 2: Comparison: Diclofenac Test (Lower Dose) vs Placebo; Test type: Superiority or Other; p = 0.091, t-test, 2 sided
Statistical Analysis 3: Comparison: Celecoxib vs Placebo; Test type: Superiority or Other; p = 0.053, t-test, 2 sided

6. Secondary Outcome: TOTPAR-8. Total Pain Relief (TOTPAR) Over 0 to 8 Hours
Description: Pain relief was assessed using a 5-point categorical scale at all assessment time points after time 0. Subjects were asked "How much relief have you had since your starting pain?" with response choices of none = 0, a little = 1, some = 2, a lot = 3, and complete = 4.
  The Total Pain Relief (TOTPAR) score for a given time interval is calculated as the sum of the pain relief scores at each follow-up time point (as recorded on the categorical pain relief scale) over that interval multiplied by the amount of time (in hours) since the prior assessment. In this way individual scores covering a longer time period were given more weight. The minimum theoretical score is 0 units, which represent no relief from pain (score of 0 on categorical scale) at all time points after time 0. The maximum theoretical score is 32 units, which represents complete relief from pain (score of 4 on a categorical scale) at all time points after time 0.
Time Frame: 0 - 8 hours
Measure: Mean (Standard Deviation); unit: units on a scale*hour
Arm/Group | Celecoxib | Diclofenac Test (Lower Dose) | Diclofenac Test (Upper Dose) | Placebo
Number analyzed (Participants) | 106 | 109 | 107 | 106
units on a scale*hour | 3.840 (6.8) | 3.690 (6.8) | 4.652 (7.5) | 1.943 (4.4)
Statistical Analysis 1: Comparison: Diclofenac Test (Upper Dose) vs Placebo; Test type: Superiority or Other; p = 0.002, t-test, 2 sided
Statistical Analysis 2: Comparison: Diclofenac Test (Lower Dose) vs Placebo; Test type: Superiority or Other; p = 0.026, t-test, 2 sided
Statistical Analysis 3: Comparison: Celecoxib vs Placebo; Test type: Superiority or Other; p = 0.017, t-test, 2 sided

7. Secondary Outcome: TOTPAR-24. Total Pain Relief (TOTPAR) Over 0 to 24 Hours
Description: Pain relief was assessed using a 5-point categorical scale at all assessment time points after time 0. Subjects were asked "How much relief have you had since your starting pain?" with response choices of none = 0, a little = 1, some = 2, a lot = 3, and complete = 4.
  The Total Pain Relief (TOTPAR) score for a given time interval is calculated as the sum of the pain relief scores at each follow-up time point (as recorded on the categorical pain relief scale) over that interval multiplied by the amount of time (in hours) since the prior assessment. In this way individual scores covering a longer time period were given more weight. The minimum theoretical score is 0 units, which represent no relief from pain (score of 0 on categorical scale) at all time points after time 0. The maximum theoretical score is 96 units, which represents complete relief from pain (score of 4 on a categorical scale) at all time points after time 0.
Time Frame: 0 - 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale*hour
Arm/Group | Celecoxib | Diclofenac Test (Lower Dose) | Diclofenac Test (Upper Dose) | Placebo
Number analyzed (Participants) | 106 | 109 | 107 | 106
units on a scale*hour | 10.670 (22.2595) | 10.186 (21.3384) | 13.325 (25.9326) | 3.566 (10.8804)
Statistical Analysis 1: Comparison: Diclofenac Test (Upper Dose) vs Placebo; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Diclofenac Test (Lower Dose) vs Placebo; Test type: Superiority or Other; p = 0.005, t-test, 2 sided
Statistical Analysis 3: Comparison: Celecoxib vs Placebo; Test type: Superiority or Other; p = 0.004, t-test, 2 sided

8. Secondary Outcome: TOTPAR-48. Total Pain Relief (TOTPAR) Over 0 to 48 Hours
Description: Pain relief was assessed using a 5-point categorical scale at all assessment time points after time 0. Subjects were asked "How much relief have you had since your starting pain?" with response choices of none = 0, a little = 1, some = 2, a lot = 3, and complete = 4.
  The Total Pain Relief (TOTPAR) score for a given time interval is calculated as the sum of the pain relief scores at each follow-up time point (as recorded on the categorical pain relief scale) over that interval multiplied by the amount of time (in hours) since the prior assessment. In this way individual scores covering a longer time period were given more weight. The minimum theoretical score is 0 units, which represent no relief from pain (score of 0 on categorical scale) at all time points after time 0. The maximum theoretical score is 192 units, which represents complete relief from pain (score of 4 on a categorical scale) at all time points after time 0.
Time Frame: 0 - 48 hours
Measure: Mean (Standard Deviation); unit: units on a scale*hour
Arm/Group | Celecoxib | Diclofenac Test (Lower Dose) | Diclofenac Test (Upper Dose) | Placebo
Number analyzed (Participants) | 106 | 109 | 107 | 106
units on a scale*hour | 22.972 (51.1) | 21.635 (48.) | 28.054 (58.1) | 4.925 (19.4)
Statistical Analysis 1: Comparison: Diclofenac Test (Upper Dose) vs Placebo; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 2: Comparison: Diclofenac Test (Lower Dose) vs Placebo; Test type: Superiority or Other; p < 0.001, t-test, 2 sided
Statistical Analysis 3: Comparison: Celecoxib vs Placebo; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Celecoxib | Diclofenac Test (Lower Dose) | Diclofenac Test (Upper Dose) | Placebo
Serious Adverse Events (participants affected / at risk) | 1/106 | 0/109 | 0/107 | 0/106
Other Adverse Events (participants affected / at risk) | 86/106 | 84/109 | 77/107 | 63/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Celecoxib (N=106) | Diclofenac Test (Lower Dose) (N=109) | Diclofenac Test (Upper Dose) (N=107) | Placebo (N=106)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Celecoxib (N=106) | Diclofenac Test (Lower Dose) (N=109) | Diclofenac Test (Upper Dose) (N=107) | Placebo (N=106)
Postprocedural edema (Injury, poisoning and procedural complications) | 35 | 36 | 35 | 34
Nausea (Gastrointestinal disorders) | 29 | 34 | 25 | 39
Headache (Nervous system disorders) | 11 | 17 | 11 | 16
Dizziness (Nervous system disorders) | 11 | 17 | 5 | 17
Vomiting (Gastrointestinal disorders) | 15 | 13 | 7 | 13
Postprocedural hematoma (Injury, poisoning and procedural complications) | 8 | 12 | 4 | 11
Constipation (Gastrointestinal disorders) | 9 | 12 | 6 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 4 | 6 | 4
Paraesthesia (Nervous system disorders) | 8 | 2 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No